CLINICAL TRIAL: NCT04549545
Title: The Vivaer® Procedure for Treatment of Nasal Airway Obstruction - A ProspecTive, Multicenter Randomized Controlled TriAl Comparing Vivaer to Sham Control (VATRAC)
Brief Title: Vivaer® Procedure for Treatment of Nasal Airway Obstruction Study
Acronym: VATRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTP1006
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Nasal Airway Obstruction
Keywords: Nasal obstruction; NAO; Nasal valve dysfunction; Nasal airway obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: 2:1 site-stratified randomization will be used to allocate participants to either the active treatment arm (Vivaer procedure) or the control arm (sham procedure). Crossover within 30 days after 3 month follow-up visit.
Who Masked: Participant
Masking Description: Participant will be blinded to the study arm they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vivaer Procedure (Active Comparator): The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session. Each side of the nose will be treated with up to four (4) non-overlapping applications of RF energy at the junction of the upper and lower lateral cartilage on the lateral nasal wall. Treatment settings to be used are: temperature 60° C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (24 months).
  Interventions: Device: Vivaer ARC Stylus
- Sham Control Procedure (Sham Comparator): The sham control procedure will be performed in the study clinic using the Vivaer ARC Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Interventions: Device: Sham

INTERVENTIONS:
Device: Vivaer ARC Stylus — The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session.
  Arms: Vivaer Procedure
Device: Sham — The sham control procedure will be performed in the study clinic using the Vivaer ARC Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Arms: Sham Control Procedure

SUMMARY:
The purpose of this study is to compare the Vivaer procedure with radiofrequency (RF) energy to sham procedure for treatment of nasal airway obstruction (NAO).

DETAILED DESCRIPTION:
The purpose of this study is to compare the Vivaer procedure for treatment of nasal airway obstruction (NAO) with a sham procedure that simulates the actual procedure as closely as possible absent the delivery of radiofrequency (RF) energy to the nasal tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years (inclusively).
2. Willing and able to provide informed consent.
3. Willing and able to comply with the subject-specific requirements outlined in the Study Protocol.
4. Seeking treatment for nasal obstruction and willing to undergo an office-based procedure.
5. Baseline Nasal Obstruction Symptom Evaluation (NOSE) Scale score ≥ 55.
6. Nasal valve is a primary or significant contributor to the patient's nasal obstruction as determined by the study investigator (based on clinical presentation, physical examination, nasal endoscopy, etc.) and the patient has a positive response to any of the following temporary measures (based on patient history or office exam):

   * Use of external nasal dilator strips (eg, Breathe Right Strips)
   * Use of internal nasal dilator cones
   * Modified Cottle Maneuver (manual elevation of the lateral nasal wall using a small instrument or cotton-tipped applicator to open the nasal valve)
   * Cottle Maneuver (manual lateral retraction of the cheek to open the nasal valve)
7. Dissatisfaction with medical management as judged by the patient. Defined as failed medical therapy (eg, decongestants, antihistamines, and/or nasal sprays for an appropriate period of time), but a positive response to internal or external nasal dilators.

Exclusion Criteria:

1. Prior surgery of the lateral nasal wall, including cephalic resection of the lower lateral cartilage, dome division or suture plication, alar graft or spreader graft placement.
2. Rhinoplasty, septoplasty, inferior turbinate reduction or functional endoscopic sinus surgery (FESS) within the preceding 3 months.
3. Severe case of any of the following: septal deviation, turbinate hypertrophy, polyps, or ptotic nose tip believed to be the primary contributor to the patient's nasal obstruction symptoms and warranting surgical intervention.
4. Any adjunctive surgical nasal procedure planned on the same day or within 6 months after the Vivaer procedure.
5. Known or suspected to be pregnant or is lactating.
6. Participating in another clinical research study.
7. Other medical conditions which in the opinion of the investigator would predispose the patient to poor wound healing or increased surgical risk, or poor compliance with the requirements of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Han, MD, Principal Investigator — EVMS Medical Group; Stacey Silvers, MD, Principal Investigator — Madison ENT
Locations (12):
- United States (12):
  - Roseville Facial Plastic Surgery, Roseville, California
  - Breathe Clear Institute, Torrance, California
  - ENT and Allergy Associates of Florida, Coral Springs, Florida
  - ENT Associates of South Florida, Fort Lauderdale, Florida
  - ENT and Allergy Associates of Florida, Port Saint Lucie, Florida
  - Advanced ENT and Allergy KY, Louisville, Kentucky
  - Madison ENT, New York, New York
  - Piedmont ENT Associates NC, Winston-Salem, North Carolina
  - Bethlehem ENT, Bethlehem, Pennsylvania
  - ENT Associates of Texas (ENTtex), McKinney, Texas
  - Ogden Clinic, Ogden, Utah
  - EVMS Ear Nose and Throat Surgeons, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silvers SL, Rosenthal JN, McDuffie CM, Yen DM, Han JK. Temperature-controlled radiofrequency device treatment of the nasal valve for nasal airway obstruction: A randomized controlled trial. Int Forum Allergy Rhinol. 2021 Dec;11(12):1676-1684. doi: 10.1002/alr.22861. Epub 2021 Jul 9. PMID 34240571
- [Result] Han JK, Silvers SL, Rosenthal JN, McDuffie CM, Yen DM. Outcomes 12 Months After Temperature-Controlled Radiofrequency Device Treatment of the Nasal Valve for Patients With Nasal Airway Obstruction. JAMA Otolaryngol Head Neck Surg. 2022 Oct 1;148(10):940-946. doi: 10.1001/jamaoto.2022.2293. PMID 36048465
- [Result] Silvers SL, McDuffie CM, Yen DM, Rosenthal JN, Davis SE, Han JK. Two-year outcomes of radiofrequency device treatment of the nasal valve for nasal airway obstruction. Rhinology. 2024 Jun 1;62(3):310-319. doi: 10.4193/RhinRhin23.377. PMID 38217847
- [Result] Han JK, Rosenthal JN, McDuffie CM, Yen DM, Bikhazi NB, Kakarlapudi VV, Silvers SL. Temperature-Controlled Radiofrequency Treatment of the Nasal Valve in Patients With Nasal Obstruction: Long-Term Outcomes. Otolaryngol Head Neck Surg. 2025 Apr;172(4):1214-1223. doi: 10.1002/ohn.1118. Epub 2025 Jan 17. PMID 39822054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Particpants were recruited based on physican referral at 16 academic medical centers and clinics between August 12,2020 and December 28, 2020. The First Participant enrolled on August 12, 2020 and the last participant enrolled on December 28, 2020.
Pre-assignment Details: There was no wash out or run in for this study
Groups:
- Active Treatment Arm: Vivaer Procedure Only: A 2:1 site-stratified randomization will be used to allocate participants with NAO to either the active treatment arm (Vivaer procedure) or the control arm (sham procedure)
  Subjects randomized to the Active Treatment will receive the Vivaer procedure.
  The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session. Each side of the nose will be treated with up to four (4) non-overlapping applications of RF energy at the junction of the upper and lower lateral cartilage on the lateral nasal wall. Treatment settings to be used are: temperature 60° C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (24 months).
  Participants in this study will undergo bilateral treatment of the nasal valves in a single study session.
  Active treatment participants (Vivaer procedure) will have an extended follow-up with evaluations conducted in-office at 6 months (26 weeks) and remotely at 12 months (52 weeks) and 24 months (104 weeks).
- Control Arm: Sham Control Procedure First, Optional Crossover to Vivaer Procedure: A 2:1 site-stratified randomization will be used to allocate participants with NAO to either the active treatment arm (Vivaer procedure) or the control arm (sham procedure)
  The sham control procedure will be performed in the study clinic using the Vivaer ARC Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Participants receiving the sham procedure may elect to crossover to the active treatment arm (Vivaer procedure) within 30 days after the 3-month follow-up evaluation provided they still meet all eligibility criteria. Continued follow-up will be conducted at 1, 3, 6, 12, and 24 months after the Vivaer procedure to provide additional information on longer-term efficacy and duration of treatment effect.
  Participants that received the sham procedure and do not elect to crossover or no longer meet all eligibility criteria will be exited from the study following the 3-month evaluation.
Period: Initial Period
Arm/Group | Active Treatment Arm: Vivaer Procedure Only | Control Arm: Sham Control Procedure First, Optional Crossover to Vivaer Procedure
Started | 78 | 41
Completed | 68 | 31
Not Completed | 10 | 10
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Additional ENT Procedure | 3 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Ineligible for Crossover and Exited as study complete | 0 | 9
Period: Crossover Period
Arm/Group | Active Treatment Arm: Vivaer Procedure Only | Control Arm: Sham Control Procedure First, Optional Crossover to Vivaer Procedure
Started | 0 (Active Treatment not eligible for Crossover) | 31
Completed | 0 (Active Treatment not eligible for Crossover) | 20
Not Completed | 0 | 11
Not completed — Additional ENT Procedure | 0 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: A total of 119 eligible patients were randomized. Assignment with 78 in the active treatment arm and 41 in the sham-control arm. One patient in the active treatment arm withdrew consent before treatment. One patient in the sham-control arm was lost to follow-up before the 3-month visit (primary endpoint).Therefore, a total of 117 patients (77 active treatment and40 sham control) were included in the analysis of the 3-month primary endpoint.
Groups:
- Active Treament Arm - Vivaer Procedure Only: The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session. Each side of the nose will be treated with up to four (4) non-overlapping applications of RF energy at the junction of the upper and lower lateral cartilage on the lateral nasal wall. Treatment settings to be used are: temperature 60° C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (24 months).
  Vivaer ARC Stylus: The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session.
- Control Sham Control Procedure First, Then Optional Crossover to Vivaer Procedure: The sham control procedure will be performed in the study clinic using the Vivaer ARC Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Sham: The sham control procedure will be performed in the study clinic using the Vivaer ARC Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
- Total: Total of all reporting groups
Arm/Group | Active Treament Arm - Vivaer Procedure Only | Control Sham Control Procedure First, Then Optional Crossover to Vivaer Procedure | Total
Number analyzed (Participants) | 78 | 41 | 119
Age, Categorical [Count of Participants; unit: Participants] — Age for inclusion 18-85 (inclusive). Age reported for overall analyzed participants
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 78 | 41 | 119
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.4) | 50.0 (11.2) | 48.5 (12.3)
Sex/Gender, Customized [Number; unit: participants] — Overall percentage for analyzed participants
  participants
    Female | 47 | 25 | 72
    Male | 30 | 15 | 45
Race/Ethnicity, Customized [Number; unit: participants] — Patients self-identified race and ethnicity. Race and ethnicity classifications were adapted from US Food and Drug Administration-recommended classifications. These data were assessed to aid in interpretation of trial generalizability and conclusions and frame any relevant implications for clinical care.
  participants
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 1 | 1 | 2
    Black or African American | 4 | 2 | 6
    White | 69 | 36 | 105
    Declined Choice | 2 | 0 | 2
Baseline NOSE Scale Score [Mean (Standard Deviation); unit: Average Score] — The primary and secondary end point measures of this trial analyzed at 3, 6, and 12 months post procedure were (1) responder rate, where a responder was defined as 20% or greater improvement (decrease) in NOSE Scale score or 1 or greater NOSE Scale severity category improvement16from baseline, and (2) the mean change in NOSE Scale score from baseline.
  Average Score | 76.7 (12.6) | 78.8 (14.3) | 77.4 (13.2)
Ease-of-breathing VAS Score [Median (Standard Deviation); unit: score] — Ease-of-breathing VAS is a 100-mm scale, where 0=no difficulty breathing and 100=extreme difficulty breathing.
  VAS=visual analog scale.
  score | 59.3 (21.6) | 61.8 (18.4) | 60.1 (20.6)

OUTCOME MEASURES:

1. Primary Outcome: Nasal Obstruction Symptom Evaluation (NOSE) Scale - 3 Month Responder Rate
Description: The Nasal Obstruction Symptom Evaluation (NOSE) Scale is a patient self-reported questionnaire consisting of 5 symptoms of nasal obstruction: nasal congestion, nasal blockage, trouble breathing, trouble sleeping, and getting enough air during exercise. Patients will report over the past 1 month how much the symptoms have been a problem. Total score ranges from 0 to 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as mild (range, 5-25), moderate (range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses.
Time Frame: 3 months visit following the study procedure.
Population: The percentage of patients designated responders, defined as 20% or greater improvement (decrease) in Nasal Obstruction Symptom Evaluation (NOSE)Scale score or 1 or greater NOSE Scale severity category improvement from baseline. Error bars indicate 95% CIs.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Active Treatment Arm: Vivaer Procedure: A 2:1 site-stratified randomization will be used to allocate participants with NAO to either the active treatment arm (Vivaer procedure) or the control arm (sham procedure)
  Subjects randomized to the Active Treatment will receive the Vivaer procedure.
  The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session. Each side of the nose will be treated with up to four (4) non-overlapping applications of RF energy at the junction of the upper and lower lateral cartilage on the lateral nasal wall. Treatment settings to be used are: temperature 60° C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (24 months).
  Participants in this study will undergo bilateral treatment of the nasal valves in a single study session.
  Active treatment participants (Vivaer procedure) will have an extended follow-up with evaluations conducted in-office at 6 months (26 weeks) and remotely at 12 months (52 weeks) and 24 months (104 weeks).
- Control Arm: Sham Control Procedure: A 2:1 site-stratified randomization will be used to allocate participants with NAO to either the active treatment arm (Vivaer procedure) or the control arm (sham procedure)
  The sham control procedure will be performed in the study clinic using the Vivaer ARC Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Participants receiving the sham procedure may elect to crossover to the active treatment arm (Vivaer procedure) within 30 days after the 3-month follow-up evaluation provided they still meet all eligibility criteria. Continued follow-up will be conducted at 1, 3, 6, 12, and 24 months after the Vivaer procedure to provide additional information on longer-term efficacy and duration of treatment effect.
  Participants that received the sham procedure and do not elect to crossover or no longer meet all eligibility criteria will be exited from the study following the 3-month evaluation.
Arm/Group | Active Treatment Arm: Vivaer Procedure | Control Arm: Sham Control Procedure
Number analyzed (Participants) | 77 | 39
percentage of participants | 88.3 [79.2 to 93.7] | 42.5 [28.5 to 57.8]

2. Secondary Outcome: Nasal Obstruction Symptom Evaluation (NOSE) Scale Mean Change From Baseline Through 3 Months
Description: The NOSE Scale is a patient self-reported questionnaire consisting of 5 symptoms of nasal obstruction: nasal congestion, nasal blockage, trouble breathing, trouble sleeping, and getting enough air during exercise. Patients will report over the past 1 month how much the symptoms have been a problem. Total score ranges from 0 to 100, where higher scores indicate worse obstruction.
  This study will measure the mean change in NOSE Scale from baseline to 3 months after procedure.
Time Frame: Change from Baseline to 3 months following the study procedure.
Population: At baseline, all patients were classified as having extreme or severe obstruction, based on the NOSE-scale severity classification system. This outcome measure shows the difference in overall score between baseline and 3 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Vivaer Procedure | Sham Control Procedure
Number analyzed (Participants) | 77 | 39
score on a scale | -42.3 [-46.6 to -37.1] | -16.8 [-26.3 to -7.2]

3. Secondary Outcome: Percentage of Participants With Treatment Related Events (Safety) - Through 3 Months
Description: Characterizing the type and frequency of adverse events reported. Subjects will be asked about possible side effects or adverse experiences related to the study procedure at each follow up visit. All events will be documented and identified as to its relationship and level of relatedness to the study device and/or study procedure. Date of onset, seriousness, intensity, duration and outcome will be documented.
Time Frame: At or following the study procedure up to to 3 months.
Population: Adverse events considered at least possibly related to the device and/or procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Vivaer Procedure | Sham Control Procedure
Number analyzed (Participants) | 77 | 39
Participants
  Vasovagal Reaction | 1 | 0
  Intermittent Nose Bleed with Mucous | 1 | 0
  Headache | 0 | 1
  No Safety Issue | 75 | 38

4. Other Pre Specified Outcome: NOSE Scale Score - 3 Month Responder Rate Improvement in NOSE Score
Description: The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of patients treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as range, 5-25), (range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  Measurement is # improvement in NOSE Scale score from baseline, the lower the score the less obstruction or a change to lower score indicates improvement in nasal airway obstruction.
  These data represents percent improvement in NOSE Scale score from baseline at 3 months
Time Frame: 3 Month
Population: The combined active treatment group contains patients from the index active treatment arm and the crossover active treatment arm. The term baseline in the index active treatment arm refers to the out-come measure value prior to original active treatment procedure, and in the case of the crossover active treatment arm, baseline refers to the value reported at the time of requalification for crossover.
Measure: Number; unit: percentage of participants
Groups:
- Combined Active Treatment (Vivaer Procedure): A total of 119 eligible patients were randomized, and 117 (77 active treatment and 40 sham control) were included in the analysis of the 3-month primary end point. After primary end point analysis and unblinding, 31 patients were eligible for crossover, and all elected to undergo active treat- ment. Two patients who crossed over were found to be ineli- gible during trial monitoring but were included in data analy- sis. Therefore, a total of 108 patients underwent active treatment in the trial.
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 107
percentage of participants | 53.6

5. Other Pre Specified Outcome: NOSE Scale Score - 3 Month Average
Description: The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of patients treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as range, 5-25), range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  These data represents the NOSE Scale average score from baseline at 3 months
Time Frame: 3 Month
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 107
score on a scale | 35.4 [30.8 to 40.1]

6. Other Pre Specified Outcome: NOSE Scale Score - 6 Month Average
Description: The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of patients treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as range, 5-25), range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  These data represents the NOSE Scale average score from baseline at 6 months
Time Frame: 6 Month
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 100
score on a scale | 33.2 [28.4 to 37.9]

7. Other Pre Specified Outcome: NOSE Scale Score - 12 Month Average
Description: The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of patients treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as range, 5-25), range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  These data represents the NOSE Scale average score from baseline at 12 months
Time Frame: 12 Month
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 88
score on a scale | 31.4 [26.3 to 36.5]

8. Other Pre Specified Outcome: NOSE Scale Score - 24 Month Average
Description: as for outcome 7
Time Frame: 24 Month
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 73
score on a scale | -41.70 [-48.80 to -34.60]

9. Other Pre Specified Outcome: NOSE Scale Score - 6 Month Responder Rate Improvement in NOSE Score
Description: The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of patients treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as range, 5-25), range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  Measurement is # improvement in NOSE Scale score from baseline
  These data represents percent improvement in NOSE Scale score from baseline at 6 months
Time Frame: 6 Month
Measure: Number; unit: percentage of participants
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 100
percentage of participants | 56.6

10. Other Pre Specified Outcome: NOSE Scale Score - 12 Month Responder Rate Improvement in NOSE Score
Description: The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of patients treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as range, 5-25), range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  These data represents percent improvement in NOSE Scale score from baseline at 12 months
Time Frame: 12 Month
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 88
percentage of participants | 58.8

11. Other Pre Specified Outcome: NOSE Scale Score -24 Month Responder Rate Improvement in NOSE Score
Description: as for outcome 10
Time Frame: 24 Month
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 73
score on a scale | 90.40 [81.50 to 95.30]

12. Other Pre Specified Outcome: Epworth Sleepiness Scale - 3 Month
Description: The ESS evaluates the self-reported likelihood of dozing or falling asleep in 8 daytime situations with likelihood rated No Chance (0), Slight (1), Moderate (2), or High Chance (3).40 The total of the scores across the 8 questions can be categorized and interpreted as: 0-7 It is unlikely that you are abnormally sleepy. 8-9 You have an average amount of daytime sleepiness. 10-15 You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention. 16-24 You are excessively sleepy and should consider seeking medical attention.
  The mean change in Epworth Sleepiness Scale score from baseline was also analyzed at 3-, 6-, and 12-months post procedure. NOSE Scale and Epworth Sleepiness Scale data were also collected at 1 month post procedure.
  Data reported here is from 3M as 12M was not included because of the long-term follow-up focus of the report.
Time Frame: 3 Months
Population: as for outcome 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 107
score on a scale | 6.5 [5.6 to 7.5]

13. Other Pre Specified Outcome: Epworth Sleepiness Scale - 6 Month
Description: as for outcome 12
Time Frame: 6 Months
Population: as for outcome 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 100
score on a scale | 6.2 [5.3 to 7.1]

14. Other Pre Specified Outcome: Epworth Sleepiness Scale - 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: as for outcome 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 88
score on a scale | 5.5 [4.6 to 6.4]

15. Other Pre Specified Outcome: Epworth Sleepiness Scale - 24 Months
Description: as for outcome 12
Time Frame: 24 Months
Population: as for outcome 4
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 73
score on a scale | 5.4 [4.5 to 6.4]

16. Other Pre Specified Outcome: Concomitant Medication and Mechanical Nasal Aid Analysis
Description: Medications tracked during the trial were antihistamines, decongestants, leukotriene inhibitors, intranasal steroids, anticholinergics, and immunotherapy. Use of nasal strips/cones was also tracked.
Time Frame: 12 Months
Measure: Number; unit: percent
Groups:
- Combined Active Treatment (Vivaer Procedure): A total of 119 eligible patients were randomized, and 117 (77 active treatment and 40 sham control) were included in the analysis of the 3-month primary end point. After primary end point analysis and unblinding, 31 patients were eligible for crossover, and all elected to undergo active treat- ment. Two patients who crossed over were found to be ineli- gible during trial monitoring but were included in data analy- sis. Therefore, a total of 108 patients underwent active treatment in the trial.
  This analysis is for 88 subjects who reached 12 month timepoint.
Arm/Group | Combined Active Treatment (Vivaer Procedure)
Number analyzed (Participants) | 88
percent
  No Change in Medication/Mechanical Aid Use | 27
  Decrease/Stopped Use in 1 Class of Medication/Mechanical Aid Use | 67
  Increase/Started 1 class of Medication/Mechanical Aid Use | 8

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Vivaer Procedure: A 2:1 site-stratified randomization will be used to allocate participants with NAO to either the active treatment arm (Vivaer procedure) or the control arm (sham procedure)
  Subjects randomized to the Active Treatment will receive the Vivaer procedure.
  The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal valves in a single study session. Each side of the nose will be treated with up to four (4) non-overlapping applications of RF energy at the junction of the upper and lower lateral cartilage on the lateral nasal wall. Treatment settings to be used are: temperature 60° C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (24 months).
  Participants in this study will undergo bilateral treatment of the nasal valves in a single study session.
  Active treatment participants (Vivaer procedure) will have an extended follow-up with evaluations conducted in-office at 6 months (26 weeks) and remotely at 12 months (52 weeks) and 24 months (104 weeks).
Arm/Group | Vivaer Procedure | Sham Control Procedure
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/39
Other Adverse Events (participants affected / at risk) | 7/108 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaer Procedure (N=108) | Sham Control Procedure (N=39)
Nasal Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Medication use was not dictated by the protocol and could affect symptom relief; Data presented are through 12 months and continued follow-up will provide additional data on long term durability. Only subjects with nasal valve collapse as primary NAO were enrolled, but some subjects may have other contributors - for this reason, eligibility exclusion criteria should be considered with results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04549545/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04549545/SAP_001.pdf